CLINICAL TRIAL: NCT03253315
Title: Clinical Audit of the Management of Pericarditis in Children.
Brief Title: Management of Pericarditis in Children.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, aya gomaa mohamed, Principal investigator, Assiut University
Other Study IDs: ayafadl24791
Record Dates: First submitted 2017-08-07; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Pericarditis
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pericardium is a double-walled sac containing the heart and the roots of the great vessels. The pericardial sac has two layers, a serous visceral l layer (also known as epicardium when it comes into contact with the myocardium) and a fibrous parietal layer. It encloses the pericardial cavity, which contains pericardial fluid. The pericardium fixes the heart to the mediastinum, gives protection against infection and provides lubrication for the heart. Pericardial diseases may be either isolated disease or part of a systemic disease Diseases of the pericardium present clinically in one of several ways

* Acute and recurrent pericarditis
* Pericardial effusion without major hemodynamic compromise
* Cardiac tamponade with cardiac compromise
* Constrictive pericarditis

DETAILED DESCRIPTION:
* Pericarditis usually present with chest pain and dyspnea. Effusion can present with no symptoms, dull ache in left chest and abdominal pain Cardiac tamponade is recognized by the excessive fall of systolic blood pressure
* Diagnostic workup A) Chest X-ray:_ chest X-ray can detect varying degree of cardiomegaly. B) Echocardiography: It is the first-line imaging test. clinically, two-dimensional echocardiography with Doppler provides the most cost-effective way of diagnosing C) Electrocardiograph D) cardiac computerized tomography :- Also may be helpful 4)Therapy of pericarditis in pediatrics the medical lines of treatment of pericarditis are:_ A)Aspirin and non-steroidal anti-inflammatory:_ are the mainstay of the therapy of inflammatory pericardial diseases B)Steroids: a minority of patients will require treatment with systemic steroid therapy as

  * Patients with symptoms refractory to standard therapy

    * Acute pericarditis due to connective tissue disease ●Uremic pericarditis C)Immunosuppressant and biological drugs (more commonly used in recurrent pericarditis) .Interventional therapeutic techniques-_

Most patients with acute pericarditis can be managed effectively with medical therapy alone. However, patients may require invasive therapies for:

* A moderate to large pericardial effusion, particularly if hemodynamically significant.
* Frequent, highly symptomatic recurrences of acute pericarditis with pericardial effusion ●Evidence of constrictive pericarditis (a late occurrence when present) A)Pericardial drainage :Prolonged catheter drainage of a pericardial effusion is an effective means of preventing fluid reaccumulation.

B)Pericardiotomy, pericardial window and pericardiectomy: pericardiectomy may be considered for frequent and highly symptomatic recurrences of pericarditis tamponade .. C)Surgical decompression of the pericardium :_can be achieved either by conventional heart surgery or video-assisted thoracoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Children with pericarditis and/or pericardial effusion above one year of age detected clinically and by echocardiography

Exclusion Criteria:

* children below one year of age. - children with malignant effusion.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients who above one year of age up to 18 years diagnosed with pericarditis and/or pericardial effusions are candidates for the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic signs | one month
  1. normal cardiac size by echocardiography (measurable by echocardiographic probe)
  2. normal thickening of pericardium by echocardiography .(measurable by echocardiographic probe)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt